CLINICAL TRIAL: NCT02657096
Title: Effectiveness of an Oral Decontaminant Agent in Addition to Non-surgical Therapy of Chronic Periodontitis: A Split Mouth Study
Brief Title: Decontaminant Agent in the Treatment of Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Dr. Gaeasno Isola, DDS,PhD Dr. Isola Gaetano, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 918-10
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Periodontitis
Keywords: Chronic Periodontitis; Hybenx; Desiccant agent; Healing; Microbiology; Periodontal Diseases; Periodontitis; Split-mouth clinical Study
MeSH Terms: conditions — Chronic Periodontitis; Periodontal Diseases; Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hybenx treatment (Experimental): Both quadrants included maxillary teeth 11-16 and 21-26. Each selected subject underwent randomly, without anaesthesia, at the same time and after recording periodontal parameters, the two following treatments: in one, maxillary quadrants were treated as conventional SRP + desiccant (Hybenx). In the maxillary quadrant assigned to SRP + hybenx treatment, hybenx was applied, after SRP, on the marginal gingiva with a 30-second incubation period and then thoroughly rinsed away through abundant irrigation with a sterile saline solution.
  Interventions: Procedure: Hybenx treatment (device); Procedure: Scaling and Root Planing (SRP)
- Scaling and Root Planing (Sham Comparator): The contra-lateral quadrants were treated as conventional Scaling and Root Planing (SRP) alone.
  Interventions: Procedure: Hybenx treatment (device); Procedure: Scaling and Root Planing (SRP)

INTERVENTIONS:
Procedure: Hybenx treatment (device) — In the maxillary quadrant assigned to SRP + hybenx treatment, hybenx was applied, after SRP, on the gingiva with a 30-second incubation period and then thoroughly rinsed away through abundant irrigation with a sterile saline solution.
Procedure: Scaling and Root Planing (SRP) — The contra-lateral quadrants were treated as conventional Scaling and Root Planing (SRP) alone.

SUMMARY:
In light of the controversy that are already approved but that however still exists regarding the efficacy and influence of the decontaminant tools for the management of Chronic Periodontitis (cp), the aim of this study was to evaluates, at 1 year follow-up, the post-treatment clinical parameters and immunological and gingival microbial profiles in patients with CP, treated by either SRP in addition to desiccant or SRP alone.

The null hypothesis to invalidate was that, after a one year follow-up, there were no variations, in relation to clinical, anti-microbial and anti-inflammatory parameters between SRP + desiccant and SRP alone treatment.

DETAILED DESCRIPTION:
This trial was conducted in accordance with the World Medical Association's Declaration of Helsinki of 1975, and reviewed in 2008. The local ethical committee of the University of Messina approved the study protocol and each patient was carefully informed about the possible inherent risks of the study and provided their informed written consent. Subjects with a diagnosis of CP (Chronic Periodontitis) were enrolled in this clinical trial.

Study design Thirty-six patients, 19 men and 17 women, aged 27 to 65 (mean age 46.7) were assessed for eligibility at the Department of Biomedical, Odontostomatological Sciences and Morphological and Functional Images at the University of Messina, Messina, Italy. This trial was conducted in agreement with the CONSORT guidelines.

In all subjects, subgingival plaque was acquired from 4 separate proximal sites at 365 days after therapy.

To permit the noninvasive specimen, all the sites chosen for analysis were isolated using cotton rolls. Subsequently, by one #40 sterilized paper point present in the commercial kit† introduced into the base of the selected site for 30 s, a subgingival plaque sample was collected.

The Gingival Crevicular Fluid (GCF) was gathered, at the same time from other four different non-contiguous interproximal sites using filter paper strips‡ as previously described. The levels of IL-1β, IL-10 and TNF-α were recognized by conventional enzyme-linked immunosorbent assay using an equation with software using a five polynomial parameter.

Each selected subject underwent randomly, without anaesthesia, at the same time and after recording periodontal parameters, the two following treatments: in one, maxillary quadrants were treated as conventional Scaling and Root Planing (SRP) + desiccant (Hybenx), while the contra-lateral quadrants were treated as conventional SRP alone.

ELIGIBILITY:
Inclusion Criteria:

1. good condition of general health,
2. a minimum of 2 teeth for each quadrant with a Pocket Depth (PD) ranging from 4-6 mm,
3. no involvement of the furcation,
4. a minimum of a six teeth per quadrant, respectively.

Exclusion Criteria:

1. periodontal therapy during the last 12 months,
2. assumption of antibiotics during the last 6 months,
3. pregnancy,
4. any systemic condition which might affect the effects of the study treatment,
5. previous or current radiation or immunosuppressive therapies,
6. use of mouthwash containing antimicrobials during the previous 3 months,
7. no use of hormonal contraceptives,
8. medication by anti-inflammatory and immunosuppressive drugs,
9. previous history of hard-drinking,
10. smoking,
11. class II and III tooth mobility.

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Probing depth (PD) | At 365 days
  Measured clinically in mm using a periodontal probe during periodontal chart

SECONDARY OUTCOMES:
Plaque and Gingival Crevicular Fluid | At 365 days
  All the sites chosen for analysis were isolated using cotton rolls. Subsequently, by one #40 sterilized paper point gently introduced into the base of the selected site for 30 s, a subgingival plaque and Gingival Crevicular Fluid sample was collected. Number of participants with treatment-related adverse events as assessed by enzyme-linked immunosorbent assay and the checkerboard DNA-DNA hybridization technique were used in order to check the secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Cordasco, DDS, Study Director — University of Messina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lombardo G, Signoretto C, Corrocher G, Pardo A, Pighi J, Rovera A, Caccuri F, Nocini PF. A topical desiccant agent in association with ultrasonic debridement in the initial treatment of chronic periodontitis: a clinical and microbiological study. New Microbiol. 2015 Jul;38(3):393-407. Epub 2015 Jul 6. PMID 26147153